CLINICAL TRIAL: NCT07199062
Title: Correlation Between Occlusal Load Distribution and Periodontal Status: A Cohort Study
Brief Title: Occlusal Load Distribution and Periodontal Status
Acronym: Perio-Occlusio
Status: Not yet recruiting | Type: Observational
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, University of Bari Aldo Moro
Other Study IDs: Perio-Uniba
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Diseases; Periodontal Pocket; Periodontitis; Periimplantitis
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Periodontitis; Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Occlusal forces are unevenly distributed among teeth during mastication, potentially predisposing certain teeth to higher functional loads. Teeth subjected to increased occlusal loading may be at greater risk of periodontal breakdown, especially in patients with pre-existing periodontal disease.

Technological advances, such as mandibular movement recording systems, allow for precise assessment of occlusal contacts and load distribution. However, the relationship between occlusal loading patterns and periodontal status remains insufficiently investigated.

This study aims to evaluate whether teeth exposed to higher masticatory loads show an association with periodontal disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years).
* Presence of natural dentition, fixed prostheses, or implant-supported fixed prostheses.
* Ability to undergo radiological (OPT) and periodontal examinations.
* Signed informed consent.

Exclusion Criteria:

* Patients wearing removable prostheses.
* Severe systemic conditions contraindicating dental treatment.
* Inability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with diagnosed periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the correlation between occlusal load distribution, recorded by mandibular movement software , and periodontal condition. | 5 months
  Sowftware analysis

SECONDARY OUTCOMES:
2. To evaluate whether teeth with higher functional loads are more frequently associated with periodontal pocketing. | 5 months
  Periodontal Chating

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Giuseppe D'Albis, Principal Investigator — University of Bari Aldo Moro; Prof. Saverio Capodiferro, Study Director — University of Bari Aldo Moro